CLINICAL TRIAL: NCT07190235
Title: The Effect of Repetitive Transcranial Magnetic Stimulation Over the Supplementary Motor Area on Gait Performance in Parkinson's Disease: A Randomized Controlled Trial
Brief Title: The Effect of rTMS Over the SMA on Gait Performance in Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20250512001
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-06

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: transcranial magnetic stimulation; Parkinson's disease; supplementary motor area; gait
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 25 Hz repetitive transcranial magnetic stimulation group (Experimental): High-frequency repetitive transcranial magnetic stimulation (25 Hz), intended to increase cortical excitability and provide facilitatory neuromodulation.
  Interventions: Device: Transcranial Magnetic Stimulation
- 1 Hz repetitive transcranial magnetic stimulation group (Experimental): Low-frequency repetitive transcranial magnetic stimulation (1 Hz), intended to decrease cortical excitability and provide inhibitory neuromodulation.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham stimulation group (Placebo Comparator): The stimulation coil is positioned identically to active TMS and emits similar auditory and scalp sensations, but delivers no significant magnetic pulse to the brain, mimicking the active intervention experience without neuromodulatory effects.
  Interventions: Device: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — The repetitive transcranial magnetic stimulation (rTMS) at different frequencies will deliver 10 sessions over 2 weeks. The participants will receive different stimulation protocols to the supplementary motor area while seated using a double-cone coil connected to a transcranial magnetic stimulator.
  Arms: 1 Hz repetitive transcranial magnetic stimulation group; 25 Hz repetitive transcranial magnetic stimulation group
Device: Transcranial Magnetic Stimulation Sham — The sham transcranial magnetic stimulation (TMS) will deliver 10 sessions over 2 weeks. The participants will receive the sham stimulation protocol to the supplementary motor area while seated using a double-cone coil connected to a transcranial magnetic stimulator.
  Arms: Sham stimulation group

SUMMARY:
This study aims to investigate the effects of high-frequency and low-frequency repetitive transcranial magnetic stimulation (rTMS) over the supplementary motor area (SMA) on gait performance, especially gait initiation, in individuals with Parkinson's disease (PD). Furthermore, the investigators will explore the impact of rTMS over the SMA on walking speed, functional mobility, and limits of stability in PD. It is hypothesized that rTMS over the SMA will improve gait performance in PD.

DETAILED DESCRIPTION:
The goal of this clinical trial is to investigate the effects of high-frequency and low-frequency rTMS over the SMA on gait performance, especially gait initiation, in individuals with PD. The primary outcome will be anticipatory postural adjustments (APAs) during gait initiation. The secondary outcome will include walking speed, the timed up-and-go test (TUG), and limits of stability.

The hypotheses are:

1. Both 25 Hz and 1 Hz rTMS will have a significant effect on gait performance, especially the gait initiation phase, as assessed by APAs in PD, compared with sham stimulation.
2. 25 Hz and 1 Hz rTMS will have a different effect on gait initiation in PD.

This study will be a three-arm, randomized, double-blind, placebo-controlled study examining the effect of 25 Hz or 1 Hz SMA-TMS compared with that observed after sham TMS. A total of 81 individuals with PD will be recruited and allocated into three different groups: 1 Hz TMS group, 25 Hz TMS group, and sham TMS group. Participants in each group will receive 10 TMS sessions over 2 weeks. Assessors will conduct evaluations at baseline, post-intervention, and 4-week post-intervention. The primary outcome will be APAs during gait initiation. The secondary outcome will include walking speed, TUG , and limits of stability.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with PD according to thecriteria set by Movement Disorder Committee,
2. with Hoehn and Yahr stages II-III, which are recognized as representing mild to moderate disease severity,
3. have self-reported difficulty in gait initiation, assessed by item 5 of the freezing of gait questionnaire (FOGQ),
4. have used a dopaminergic medication dose in the last month,
5. a minimum score of 23 of 30 points on the Montreal Cognitive Assessment (MoCA).

Exclusion Criteria:

1. patients with unstable medical conditions,
2. unable to provide informed consent,
3. other neurological conditions including stroke,
4. contraindications for TMS,
5. experienced deep brain stimulation treatment,
6. no recordable motor evoked potentials (MEPs) with TMS.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2026-01-06 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in duration of anticipatory postural adjustments (APAs) during gait initiation | Baseline, 2 weeks (post-intervention)
  The duration of APAs will be calculated from the center of pressure displacement trajectory, recorded by a force plate and Vicon motion capture system.

SECONDARY OUTCOMES:
Change in duration of anticipatory postural adjustments (APAs) during gait initiation | Baseline and 6 weeks (4-week post-intervention)
  The duration of APAs will be calculated from the center of pressure displacement trajectory, recorded by a force plate and Vicon motion capture system.
Change in comfortable walking speed of the 10-meter walk test | Baseline, 2 weeks (post-intervention), 6 weeks (4-week post-intervention)
  Comfortable walking speed is a critical outcome due to its reliability, sensitivity to change, and clinical relevance in reflecting functional mobility and disease progression. This study will use 10-meter walk test to measure the walking speed.
Change in fast walking speed of the 10-meter walk test | Baseline, 2 weeks (post-intervention), 6 weeks (4-week post-intervention)
  Fast gait speed was assessed by taking an average of three trials of a 10-meter walk test (as fast as one can safely walk). Walking at high speeds poses a challenge for individuals with PD, as bradykinesia, while fast walking demands greater balance and postural stability. Fast gait speed has excellent test-retest reliability with an intraclass correlation coefficient (ICC) of 0.97 in individuals with PD.
Changes in Timed Up-and-Go Test (TUG) | Baseline, 2 weeks (post-intervention), 6 weeks (4-week post-intervention)
  The TUG is a reliable and valid test used to assess functional mobility and walking capacity in PD and requires the individual to stand up from a chair, walk seven meters, turn around, walk back to the chair, and sit down. The time taken to complete the task is recorded, with longer times indicating poorer mobility. It is commonly used in geriatric populations to evaluate fall risk and in individuals with various health conditions, including PD.
Change in Unified Parkinson's Disease Rating Scale-motor examination (UPDRS-III) | Baseline, 2 weeks (post-intervention), 6 weeks (4-week post-intervention)
  UPDRS-III is used to assess motor symptoms in PD. It is a scale with 33 scores based on 18 questions with several right, left, or other body distribution scores. It evaluates motor symptoms such as tremor, rigidity, bradykinesia, postural instability, and gait. All items have 5 response options with uniform anchors of normal rated 0, slight rated 1, mild rated 2, moderate rated 3, and severe rated 4. Higher scores indicate greater impact of PD symptoms, providing a comprehensive overview of motor abilities and aiding in the monitoring of disease progression and treatment efficacy.
Change in score of Mini-Balance Evaluation System Test (MiniBEST) | Baseline, 2 weeks (post-intervention), 6 weeks (4-week post-intervention)
  The Mini-BEST is a clinical tool designed to assess balance in individuals with PD and other conditions. It evaluates dynamic balance, functional mobility, sensory organization, APAs, postural responses, and dynamic gait. The test consists of 14 items and is scored out of 28 points, with uniform anchors of normal rated 0, moderate rated 1, and severe rated 2.
Change in freezing of gait questionnaire (FOGQ) | Baseline, 2 weeks (post-intervention), 6 weeks (4-week post-intervention)
  The FOGQ is a self-report questionnaire specifically designed to evaluate the presence and severity of FOG in patients with PD. FOG is a phenomenon where patients temporarily feel as though their feet are glued to the floor, impeding their ability to walk. The FOGQ helps in quantifying the impact of FOG on daily living and can guide therapeutic interventions. This questionnaire comprised six questions (maximum score 24 points) that sought to assess both freezing of gait, as well as gait disturbance.
Change in the 39-item Parkinson's disease questionnaire (PDQ-39) | Baseline, 2 weeks (post-intervention), 6 weeks (4-week post-intervention)
  PDQ-39 is a widely used tool to assess the health-related quality of life in individuals with PD. It consists of 39 questions that cover various aspects of daily living, including mobility, emotional well-being, social support, and activities of daily living. The PDQ-39 is designed to capture both physical and psychological impacts of the disease, helping clinicians evaluate the extent to which Parkinson's disease affects a patient's quality of life.
Change in resting motor threshold (RMT) | Baseline, 2 weeks (post-intervention), 6 weeks (4-week post-intervention)
  The RMT is the minimum stimulus intensity that evokes responses of approximately 100 µV with a similar shape and latency in 5 out of 10 successive stimuli.
Change in short-interval intracortical inhibition (SICI) | Baseline, 2 weeks (post-intervention), 6 weeks (4-week post-intervention)
  SICI is the measure of the intracortical inhibition mediated by GABAA receptors.
Intracortical facilitation (ICF) | Baseline, 2 weeks (post-intervention), 6 weeks (4-week post-intervention)
  ICF is the measure of the intracortical facilitation mediated by glutamate receptors.
Changes in the slope of the stimulus response curve (SRC) | Baseline, 2 weeks (post-intervention), 6 weeks (4-week post-intervention)
  The Changes in the slope of the stimulus-response curve (SRC) as an outcome measure refer to how the steepness of the SRC varies, reflecting the rate at which the motor evoked potential (MEP) amplitude increases in response to increasing stimulus intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Kowloon, Hong Kong

REFERENCES:
- [Background] Rahimpour S, Rajkumar S, Hallett M. The Supplementary Motor Complex in Parkinson's Disease. J Mov Disord. 2022 Jan;15(1):21-32. doi: 10.14802/jmd.21075. Epub 2021 Nov 25. PMID 34814237
- [Background] Mi TM, Garg S, Ba F, Liu AP, Wu T, Gao LL, Dan XJ, Chan P, McKeown MJ. High-frequency rTMS over the supplementary motor area improves freezing of gait in Parkinson's disease: a randomized controlled trial. Parkinsonism Relat Disord. 2019 Nov;68:85-90. doi: 10.1016/j.parkreldis.2019.10.009. Epub 2019 Oct 11. PMID 31689588
- [Background] Jacobs JV, Lou JS, Kraakevik JA, Horak FB. The supplementary motor area contributes to the timing of the anticipatory postural adjustment during step initiation in participants with and without Parkinson's disease. Neuroscience. 2009 Dec 1;164(2):877-85. doi: 10.1016/j.neuroscience.2009.08.002. Epub 2009 Aug 7. PMID 19665521
- [Background] Delval A, Tard C, Defebvre L. Why we should study gait initiation in Parkinson's disease. Neurophysiol Clin. 2014 Jan;44(1):69-76. doi: 10.1016/j.neucli.2013.10.127. Epub 2013 Oct 30. PMID 24502907
- [Background] Chen Y, Jiang H, Wei Y, Ye S, Jiang J, Mak MKY, Pang MYC, Gao Q, Huang M. Effects of non-invasive brain stimulation over the supplementary motor area on motor function in Parkinson's disease: A systematic review and meta-analysis. Brain Stimul. 2025 Jan-Feb;18(1):1-14. doi: 10.1016/j.brs.2024.12.005. Epub 2024 Dec 11. PMID 39667490
- [Background] Armstrong MJ, Okun MS. Diagnosis and Treatment of Parkinson Disease: A Review. JAMA. 2020 Feb 11;323(6):548-560. doi: 10.1001/jama.2019.22360. PMID 32044947